CLINICAL TRIAL: NCT01137097
Title: Value of Sentinel Lymph Node Biopsy to Lateral Neck Lymph Node in Thyroid Carcinoma: Prospective Study
Brief Title: Lateral Neck Sentinel Lymph Node Biopsy(LSLNB)in PTC
Acronym: LSLNB
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jee soo Kim, Association professor, Samsung Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-07-101
Record Dates: First submitted 2010-06-02; First posted 2010-06-04 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Thyroid Neoplasm
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lateral sentinel group (Active Comparator): Lateral sentinel lymph node biopsy with radioisotope
  Interventions: Procedure: Lateral sentinel lymph node biopsy
- No intervention for lateral neck (No Intervention): No lateral sentinel lymph node biopsy with radioisotope

INTERVENTIONS:
Procedure: Lateral sentinel lymph node biopsy — Sentinel lymph node biopsy with radioisotope. Isotope injection and lymphoscintigraphy preoperatively
  Arms: Lateral sentinel group

SUMMARY:
Objective: To investigate the incidence of lateral neck node occult metastasis and to show the usefulness of sentinel lymph node biopsy (SLNB) in the detection of lateral neck node metastasis in thyroid carcinoma, the investigators used a radioisotope to detect the sentinel lymph node.

Summary Background Data: Although occult lymph node metastasis to the lateral neck compartment is common in papillary thyroid carcinoma, the incidence and patterns of lateral neck node metastasis in papillary carcinoma are not known.

DETAILED DESCRIPTION:
On the day of the operation, patients underwent preoperative lymphoscintigraphy after the intratumoral injection of a Tc-99m phytate 1 mCi in 0.1-0.2 mL 0.9% NaCl under ultrasonographic guidance. Total thyroidectomy or lobectomy with central neck dissection preceded SLN detection to avoid interference by primary tumor radioactivity. After total thyroidectomy or lobectomy, the dissections were performed toward the internal jugular chain beneath the sternocleidomastoid muscle. A handheld, collimated gamma probe and lymphoscintigraphy were used to scan the lateral compartments (through skin and under the SCM) for "radioactive" lymph nodes. Removed SLNs were submitted immediately for frozen biopsy. If any of the SLNs were positive for metastasis on the frozen sections, MRND was performed immediately. In cases for which the frozen section was negative but the final pathology report detailed microscopic positivity in the lateral sentinel nodes, RAI ablations were performed without additional MRND.

ELIGIBILITY:
Inclusion Criteria:

* Cases with tumors larger than 1 cm in size or with suspicious central neck node metastasis in Papillary thyroid cancer

Exclusion Criteria:

* The patient with definite metastatic lymph node in lateral neck compartment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2009-06; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
The usefulness of lateral sentinel lymph node biopsy in PTC | at Oct 2011

CONTACTS AND LOCATIONS:
Overall Officials: Se Kyung Lee, M.D, Study Director — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No